CLINICAL TRIAL: NCT03315130
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of RA101495 in Subjects With Generalized Myasthenia Gravis
Brief Title: Safety and Efficacy Study of RA101495 in Subjects With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA101495-02.201
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.1 mg/kg zilucoplan (RA101495) (Experimental)
  Interventions: Drug: zilucoplan (RA101495)
- 0.3 mg/kg zilucoplan (RA101495) (Experimental)
  Interventions: Drug: zilucoplan (RA101495)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zilucoplan (RA101495) — Daily subcutaneous (SC) injection
  Arms: 0.1 mg/kg zilucoplan (RA101495); 0.3 mg/kg zilucoplan (RA101495)
Drug: Placebo — Daily subcutaneous (SC) injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of RA101495 in patients with generalized Myasthenia Gravis (gMG). Subjects will be randomized in a 1:1:1 ratio to receive daily SC doses of 0.1 mg/kg RA101495, 0.3 mg/kg RA101495, or matching placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gMG [Myasthenia Gravis Foundation of America (MGFA) Class II-IVa] at Screening
* Positive serology for acetylcholine receptor (AChR) autoantibodies
* QMG score ≥ 12 at Screening and Randomization
* No change in corticosteroid dose for at least 30 days prior to Randomization or anticipated to occur during the 12-week Treatment Period
* No change in immunosuppressive therapy, including dose, for at least 30 days prior to Randomization or anticipated to occur during the 12-week Treatment Period

Exclusion Criteria:

* Thymectomy within 6 months prior to Randomization or scheduled to occur during the 12 week Treatment Period
* History of meningococcal disease
* Current or recent systemic infection within 2 weeks prior to Randomization or infection requiring intravenous (IV) antibiotics within 4 weeks prior to Randomization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (30):
- United States (26):
  - Diagnostic and Medical Clinic - Mobile, Mobile, Alabama
  - The Research Center of Southern California, Carlsbad, California
  - UCLA Medical Center, Los Angeles, California
  - University of California Irvine Health ALS and Neuromuscular Center, Orange, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - University of Buffalo, Buffalo, New York
  - Hospital for Special Surgery, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Allegheny Neurological Associates, Pittsburgh, Pennsylvania
  - Wesley Neurology Clinic, Cordova, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Center for Neurological Disorders, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre University Hospital, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Howard JF Jr, Nowak RJ, Wolfe GI, Freimer ML, Vu TH, Hinton JL, Benatar M, Duda PW, MacDougall JE, Farzaneh-Far R, Kaminski HJ; Zilucoplan MG Study Group; Barohn R, Dimachkie M, Pasnoor M, Farmakidis C, Liu T, Colgan S, Benatar MG, Bertorini T, Pillai R, Henegar R, Bromberg M, Gibson S, Janecki T, Freimer M, Elsheikh B, Matisak P, Genge A, Guidon A, David W, Habib AA, Mathew V, Mozaffar T, Hinton JL, Hewitt W, Barnett D, Sullivan P, Ho D, Howard JF Jr, Traub RE, Chopra M, Kaminski HJ, Aly R, Bayat E, Abu-Rub M, Khan S, Lange D, Holzberg S, Khatri B, Lindman E, Olapo T, Sershon LM, Lisak RP, Bernitsas E, Jia K, Malik R, Lewis-Collins TD, Nicolle M, Nowak RJ, Sharma A, Roy B, Nye J, Pulley M, Berger A, Shabbir Y, Sachdev A, Patterson K, Siddiqi Z, Sivak M, Bratton J, Small G, Kohli A, Fetter M, Vu T, Lam L, Harvey B, Wolfe GI, Silvestri N, Patrick K, Zakalik K, Duda PW, MacDougall J, Farzaneh-Far R, Pontius A, Hoarty M. Clinical Effects of the Self-administered Subcutaneous Complement Inhibitor Zilucoplan in Patients With Moderate to Severe Generalized Myasthenia Gravis: Results of a Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Trial. JAMA Neurol. 2020 May 1;77(5):582-592. doi: 10.1001/jamaneurol.2019.5125. PMID 32065623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in October 2017 and concluded in November 2020.
Pre-assignment Details: The Participant flow refers to the Intent-to-treat Set for the main portion and Safety Set for the extension portion.
Groups:
- RA101495 0.1 mg/kg: Participants received RA101495 0.1 milligram/kilogram (mg/kg) as a subcutaneous injection once daily for 12 weeks in the main portion. Participants who completed main portion and were eligible to enter in the extension portion, continued receiving RA101495 0.1 mg/kg up to 48 weeks (until protocol amendment v3.0) in the extension portion (EP).
- RA101495 0.3 mg/kg: Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. At the end of the treatment period in the main portion, participants received the same dose of study drug in the extension portion until RA101495 is approved and available in the territory, or the sponsor terminates development of RA101495 for generalized myasthenia gravis (gMG). In countries where RA101495 is not approved or marketed, but in which sponsored clinical studies had been conducted, participants received RA101495 through a compassionate use pathway in the extension portion (up to 122 weeks).
- Placebo: Participants received placebo matched to RA101495 as a subcutaneous injection once daily for 12 weeks in the main portion. At the end of the treatment period in the main portion, participants were randomized to receive either RA101495 0.1 mg/kg (up to 48 weeks) or RA101495 0.3 mg/kg (up to 122 weeks) in the extension portion, as a subcutaneous injection once daily.
- RA101495 0.1 mg/kg (Before Switch) to 0.3 mg/kg (After Switch): Following implementation of protocol amendment v3.0, and upon appropriate reconsent, all study participants ongoing in the extension portion who had previously received the RA101495 0.1mg/kg/day dose switched to receive the RA101495 0.3mg/kg/day until RA101495 is approved and available in the territory, or the sponsor terminates development of RA101495 for gMG. In countries where RA101495 is not approved or marketed, but in which sponsored clinical studies had been conducted, participants received RA101495 through a compassionate use pathway in the extension portion (up to 122 weeks).
Period: Main Portion (12 Weeks)
Arm/Group | RA101495 0.1 mg/kg | RA101495 0.3 mg/kg | Placebo | RA101495 0.1 mg/kg (Before Switch) to 0.3 mg/kg (After Switch)
Started | 15 | 15 | 15 | 0
Completed | 15 | 13 | 15 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Subject withdrew consent | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: EP:Before Switch to 0.3 mg/kg(Week13-48)
Arm/Group | RA101495 0.1 mg/kg | RA101495 0.3 mg/kg | Placebo | RA101495 0.1 mg/kg (Before Switch) to 0.3 mg/kg (After Switch)
Started | 22 ((15 [who received RA101495 0.1 mg/kg] + 7 [crossover from placebo])) | 21 ((14 [who received RA101495 0.3 mg/kg + 7 [crossover from placebo] + 1 [Subject who withdrew consent in Main Portion rejoined])) | 0 | 0
Completed | 21 | 21 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Subject withdrew consent | 1 | 0 | 0 | 0
Period: EP:After Switch to 0.3 mg/kg(Week48-122)
Arm/Group | RA101495 0.1 mg/kg | RA101495 0.3 mg/kg | Placebo | RA101495 0.1 mg/kg (Before Switch) to 0.3 mg/kg (After Switch)
Started | 0 | 21 | 0 | 21
Completed | 0 | 17 | 0 | 20
Not Completed | 0 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Subject withdrew consent | 0 | 1 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- RA101495 0.1 mg/kg: Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants who completed main portion and were eligible to enter in the extension period, continued receiving RA101495 0.1 mg/kg up to 48 weeks (until protocol amendment v3.0) in the extension portion.
- Total: Total of all reporting groups
Arm/Group | RA101495 0.1 mg/kg | RA101495 0.3 mg/kg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 13 | 38
  >=65 years | 1 | 4 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (15.6) | 54.5 (14.9) | 48.4 (15.7) | 49.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 11 | 24
  Male | 7 | 10 | 4 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 2
  Black or African American | 2 | 3 | 2 | 7
  White | 13 | 11 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Main Portion: Change From Baseline to Week 12 in Quantitative Myasthenia Gravis (QMG) Score
Description: The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for myasthenia gravis (MG). The scale consists of 13 individual assessments, each scored on a 0-3 point scale (i.e., 0=none, 1=mild, 2=moderate, and 3=severe). The total score is the sum of the individual scores with a range of 0-39. Higher scores are representative of more severe impairment.
Time Frame: From Baseline to Week 12
Population: The modified ITT (mITT) population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- RA101495 0.1 mg/kg (mITT): Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the mITT population which included all participants in the ITT population who had received at least 1 dose of study drug.
- RA101495 0.3 mg/kg (mITT): Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the mITT population which included all participants in the ITT population who had received at least 1 dose of study drug.
- Placebo (mITT): Participants received placebo matched to RA101495 as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the mITT population which included all participants in the ITT population who had received at least 1 dose of study drug.
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | -5.5 (1.2) | -6.0 (1.2) | -3.2 (1.2)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0941, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -2.3, 80% CI 2-sided [-4.5 to -0.1], Standard Error of Mean 1.7 — LS mean difference and associated confidence interval are presented for each active treatment arm compared to the Placebo treatment arm
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0538, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -2.8, 80% CI 2-sided [-5.1 to -0.6], Standard Error of Mean 1.7 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Main Portion: Change From Baseline to Week 12 in the Myasthenia Gravis - Activities of Daily Living (MG-ADL) Scale
Description: The MG-ADL is a brief 8-item survey designed to evaluate MG symptom severity. The scale consists of 8 items each scored on a 0-3 point scale (i.e., 0=none, 1=mild, 2=moderate, and 3=severe). The total score is the sum of the 8 individual scores with range of 0-24. Higher scores are associated with more severe symptoms of MG.
Time Frame: From Baseline to Week 12
Population: The mITT population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | -3.3 (0.9) | -3.4 (0.9) | -1.1 (0.9)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0470, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -2.2, 80% CI 2-sided [-3.9 to -0.5], Standard Error of Mean 1.3 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0392, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -2.3, 80% CI 2-sided [-4.0 to -0.6], Standard Error of Mean 1.3 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Main Portion: Change From Baseline to Week 12 in the Myasthenia Gravis - Quality of Life 15r (MG-QOL15r) Survey
Description: The MG-QOL15r is a 15-item survey that was designed to assess quality of life in participants with MG. The survey consisted of 15 questions and the corresponding responses were each scored on a 0-2 point scale (0=Not much at all, 1=Somewhat, 2=Very Much). The total score is the sum of the 15 individual item scores with a range of 0-30. Higher scores indicate more severe impact of the disease on aspects of the participant's life.
Time Frame: From Baseline to Week 12
Population: The mITT population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | -7.4 (1.7) | -5.9 (1.7) | -2.1 (1.7)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0170, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -5.3, 80% CI 2-sided [-8.4 to -2.1], Standard Error of Mean 2.4 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0624, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -3.7, 80% CI 2-sided [-6.9 to -0.6], Standard Error of Mean 2.4 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Main Portion: Change From Baseline to Week 12 in the MG Composite Scale Total Score
Description: The MG Composite is a 10-item scale that has been used to measure the clinical status of participants with MG, in order to evaluate treatment response. It consists of 10 items which included ptosis (score range=0 to 3), double vision on lateral gaze left/right/both (score range=0 to 4), eye closure (score range=0 to 2), talking (score range=0 to 6), chewing (score range=0 to 6), swallowing (score range=0 to 6), breathing (score range=0 to 9), neck flexion or extension (score range=0 to 4), shoulder abduction (score range=0 to 5) and hip flexion (score range= 0 to 5). The total score is the sum of the 10 individual scores with a range of 0-50. Higher scores in the MG Composite indicate more severe impairment due to the disease.
Time Frame: From Baseline to Week 12
Population: The mITT population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | -5.3 (1.5) | -7.4 (1.6) | -3.3 (1.6)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.1866, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -2.0, 80% CI 2-sided [-4.9 to 0.9], Standard Error of Mean 2.2 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (mITT) vs Placebo (mITT); Test type: Superiority; p = 0.0391, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -4.1, 80% CI 2-sided [-7.0 to -1.1], Standard Error of Mean 2.2 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Main Portion: Percentage of Participants With >= 3-point Reduction in QMG Total Score at Week 12
Description: The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The scale consists of 13 individual assessments, each scored on a 0-3 point scale (i.e., 0=none, 1=mild, 2=moderate, and 3=severe). The total score is the sum of the individual scores with a range of 0-39. Higher scores are representative of more severe impairment.
Time Frame: Week 12
Population: The mITT population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
percentage of participants | 66.7 | 71.4 | 53.3

6. Secondary Outcome: Main Portion: Percentage of Participants Who Required Rescue Therapy Over the 12-week Treatment Period
Description: Percentage of participants who used at least 1 dose of rescue medication were reported.
Time Frame: Up to Week 12
Population: The mITT population included all participants in the ITT population who had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | RA101495 0.1 mg/kg (mITT) | RA101495 0.3 mg/kg (mITT) | Placebo (mITT)
Number analyzed (Participants) | 15 | 14 | 15
percentage of participants | 6.7 | 0 | 20.0

7. Secondary Outcome: Main Portion: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulted in death, life-threatening, significant or persistent disability/incapacity, congenital anomaly/birth defect, important medical event, initial inpatient hospitalization or prolongation of hospitalization.
Time Frame: From Baseline to Week 12
Population: The safety population included all participants who had received at least 1 dose of study drug (i.e., mITT Population), with participants to be analyzed based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- RA101495 0.1 mg/kg (SS): Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the safety set (SS) population which included all participants who had received at least 1 dose of study drug (i.e., mITT Population), with participants to be analyzed based on the actual treatment received.
- RA101495 0.3 mg/kg (SS): Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the SS population which included all participants who had received at least 1 dose of study drug (i.e., mITT Population), with participants to be analyzed based on the actual treatment received.
- Placebo (SS): Participants received placebo matched to RA101495 as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the SS population which included all participants who had received at least 1 dose of study drug (i.e., mITT Population), with participants to be analyzed based on the actual treatment received.
Arm/Group | RA101495 0.1 mg/kg (SS) | RA101495 0.3 mg/kg (SS) | Placebo (SS)
Number analyzed (Participants) | 15 | 14 | 15
Participants
  AEs | 15 | 12 | 14
  SAEs | 0 | 5 | 3

8. Secondary Outcome: Main Portion: Change From Baseline in Sheep Red Blood Cell (sRBC) Lysis Assay at Week 12 (Pre-dose)
Description: A BioTek ELx800 automated microplate reader is used to measure the optical density at 415 nanometer (nm) of human plasma samples to calculate the percent lysis of sheep erythrocytes that has occurred as a result of total complement activity. The measure of complement activity is determined by the degree of hemolysis of the erythrocytes.
Time Frame: Baseline and Week 12 (Pre-dose)
Population: The pharmacodynamic (PD) population included all participants in mITT Population who had at least 1 evaluable PD assessment.
Measure: Least Squares Mean (Standard Error); unit: percent lysis of sheep erythrocytes
Groups:
- RA101495 0.1 mg/kg (PD): Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed PD population which included all participants in mITT population who had at least 1 evaluable PD assessment.
- RA101495 0.3 mg/kg (PD): Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed PD population which included all participants in mITT population who had at least 1 evaluable PD assessment.
- Placebo (PD): Participants received placebo matched to RA101495 as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed PD population which included all participants in mITT population who had at least 1 evaluable PD assessment.
Arm/Group | RA101495 0.1 mg/kg (PD) | RA101495 0.3 mg/kg (PD) | Placebo (PD)
Number analyzed (Participants) | 15 | 14 | 15
percent lysis of sheep erythrocytes | -81.822 (2.469) | -94.914 (2.908) | 0.775 (2.571)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (PD) vs Placebo (PD); Test type: Superiority; p < 0.0001, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -82.597, 80% CI 2-sided [-87.249 to -77.946], Standard Error of Mean 3.563 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (PD) vs Placebo (PD); Test type: Superiority; p < 0.0001, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = -95.689, 80% CI 2-sided [-100.794 to -90.585], Standard Error of Mean 3.910 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Main Portion: Change From Baseline in C5 Levels at Week 12 (Pre-dose)
Description: Blood samples were collected from participants to assess Complement Component 5C levels.
Time Frame: Baseline and Week 12 (Pre-dose)
Population: The PD population included all participants in mITT Population who had at least 1 evaluable PD assessment.
Measure: Least Squares Mean (Standard Error); unit: micrograms/milliliter (ug/mL)
Groups:
- RA101495 0.3 mg/kg (PD): Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in main portion. Participants formed PD population which included all participants in mITT population who had at least 1 evaluable PD assessment.
Arm/Group | RA101495 0.1 mg/kg (PD) | RA101495 0.3 mg/kg (PD) | Placebo (PD)
Number analyzed (Participants) | 15 | 14 | 15
micrograms/milliliter (ug/mL) | 57.349 (7.057) | 54.302 (6.804) | -2.774 (6.237)
Statistical Analysis 1: Comparison: RA101495 0.1 mg/kg (PD) vs Placebo (PD); Test type: Superiority; p < 0.0001, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = 60.123, 80% CI 2-sided [47.839 to 72.408], Standard Error of Mean 9.394 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: RA101495 0.3 mg/kg (PD) vs Placebo (PD); Test type: Superiority; p < 0.0001, ANCOVA — 1-sided p-value is presented for each active treatment arm compared to the Placebo treatment arm; LS Mean Difference = 57.076, 80% CI 2-sided [44.955 to 69.197], Standard Error of Mean 9.269 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Main Portion: Plasma Concentration of RA101495 and Its Major Metabolites
Description: RA102758 and RA103488 are the metabolites of RA101495.
Time Frame: 1, 3 and 6 hours postdose on Day 1; Pre-dose on Week 1, 2, 4, 8 and 12
Population: The pharmacokinetic (PK) population included all participants in mITT population who had at least 1 evaluable PK assessment. Here "Number Analyzed" signifies number of participants who were evaluable at specified time points. 1 Participant (who was randomized to Placebo) mistakenly received Zilucoplan on Day 1 following a dispensing error (which was documented as a minor PD). Due to data confidentiality reasons, the results have not been reported for the placebo arm.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Groups:
- RA101495 0.1 mg/kg (PK): Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the PK population which included all participants in mITT population who had at least 1 evaluable PK assessment.
- RA101495 0.3 mg/kg (PK): Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants formed the PK population which included all participants in mITT population who had at least 1 evaluable PK assessment.
Arm/Group | RA101495 0.1 mg/kg (PK) | RA101495 0.3 mg/kg (PK)
Number analyzed (Participants) | 15 | 14
nanograms/milliliter (ng/mL)
  RA101495- Day 1: 1 hour postdose: number analyzed (Participants) | 14 | 14
  RA101495- Day 1: 1 hour postdose | 652.136 (354.652) | 2272.257 (1246.128)
  RA101495- Day 1: 3 hours postdose | 1691.267 (469.766) | 4176.000 (1211.166)
  RA101495- Day 1: 6 hours postdose: number analyzed (Participants) | 14 | 13
  RA101495- Day 1: 6 hours postdose | 1925.357 (330.335) | 4636.000 (809.804)
  RA101495- Week 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA101495- Week 1: Pre-dose | 4571.214 (719.566) | 9223.786 (2365.168)
  RA101495- Week 2: Pre-dose: number analyzed (Participants) | 15 | 13
  RA101495- Week 2: Pre-dose | 4914.200 (743.215) | 10222.846 (1662.869)
  RA101495- Week 4: Pre-dose: number analyzed (Participants) | 14 | 12
  RA101495- Week 4: Pre-dose | 5100.286 (859.767) | 10265.917 (1604.004)
  RA101495- Week 8: Pre-dose: number analyzed (Participants) | 15 | 12
  RA101495- Week 8: Pre-dose | 5222.067 (688.427) | 10075.000 (1872.400)
  RA101495- Week 12: Pre-dose: number analyzed (Participants) | 15 | 13
  RA101495- Week 12: Pre-dose | 5281.333 (1122.372) | 10284.846 (1771.586)
  RA102758- Day 1: 1 hour postdose: number analyzed (Participants) | 14 | 14
  RA102758- Day 1: 1 hour postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above lower limit of quantification (LLOQ). | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA102758- Day 1: 3 hours postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA102758- Day 1: 6 hours postdose: number analyzed (Participants) | 14 | 13
  RA102758- Day 1: 6 hours postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA102758- Week 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA102758- Week 1: Pre-dose | 252.693 (78.909) | 849.743 (273.388)
  RA102758- Week 2: Pre-dose: number analyzed (Participants) | 15 | 13
  RA102758- Week 2: Pre-dose | 408.847 (94.773) | 1473.431 (440.496)
  RA102758- Week 4: Pre-dose: number analyzed (Participants) | 14 | 12
  RA102758- Week 4: Pre-dose | 462.486 (180.098) | 1567.692 (557.745)
  RA102758- Week 8: Pre-dose: number analyzed (Participants) | 15 | 12
  RA102758- Week 8: Pre-dose | 474.073 (157.549) | 1432.808 (530.377)
  RA102758- Week 12: Pre-dose: number analyzed (Participants) | 15 | 13
  RA102758- Week 12: Pre-dose | 465.665 (195.227) | 1459.062 (451.013)
  RA103488- Day 1: 1 hour postdose: number analyzed (Participants) | 14 | 14
  RA103488- Day 1: 1 hour postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA103488- Day 1: 3 hours postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA103488- Day 1: 6 hours postdose: number analyzed (Participants) | 14 | 13
  RA103488- Day 1: 6 hours postdose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | 85.832 (257.664)
  RA103488- Week 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA103488- Week 1: Pre-dose | 356.186 (162.209) | 838.907 (255.419)
  RA103488- Week 2: Pre-dose: number analyzed (Participants) | 15 | 13
  RA103488- Week 2: Pre-dose | 501.847 (218.467) | 1135.731 (270.004)
  RA103488- Week 4: Pre-dose: number analyzed (Participants) | 14 | 12
  RA103488- Week 4: Pre-dose | 536.266 (275.013) | 1191.783 (251.853)
  RA103488- Week 8: Pre-dose: number analyzed (Participants) | 15 | 12
  RA103488- Week 8: Pre-dose | 615.740 (229.359) | 1234.708 (201.055)
  RA103488- Week 12: Pre-dose: number analyzed (Participants) | 15 | 13
  RA103488- Week 12: Pre-dose | 621.813 (241.354) | 1307.492 (331.553)

11. Secondary Outcome: Main Portion: Maximum Plasma Concentration (Cmax) on Day 1
Description: Cmax is defined as the maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 3 and 6 hours postdose on Day 1
Population: The PK Population included all participants in mITT population who had at least 1 evaluable PK assessment. 1 Participant (who was randomized to Placebo) mistakenly received Zilucoplan on Day 1 following a dispensing error (which was documented as a minor PD). Due to data confidentiality reasons, the results have not been reported for the placebo arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RA101495 0.1 mg/kg (PK) | RA101495 0.3 mg/kg (PK)
Number analyzed (Participants) | 15 | 14
ng/mL | 1945.467 (407.273) | 4858.643 (1004.457)

12. Secondary Outcome: Main Portion: Time Corresponding to Cmax (Tmax) on Day 1
Description: Tmax is defined as the time to observe maximum plasma concentration.
Time Frame: Pre-dose, 1, 3 and 6 hours postdose on Day 1
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | RA101495 0.1 mg/kg (PK) | RA101495 0.3 mg/kg (PK)
Number analyzed (Participants) | 15 | 14
hours | 4.550 [2.95 to 5.50] | 4.700 [2.62 to 5.92]

13. Secondary Outcome: Main Portion: Metabolites (RA102758 and RA103488) to Parent Ratio
Description: RA102758 and RA103488 are the metabolites of RA101495.
Time Frame: Pre-dose, 1, 3 and 6 hours postdose on Day 1; Pre-dose on Week 1, 2, 4, 8 and 12
Population: The PK Population included all participants in mITT population who had at least 1 evaluable PK assessment. Here "Number Analyzed" signifies number of participants who were evaluable at specified time points. 1 Participant (who was randomized to Placebo) mistakenly received Zilucoplan on Day 1 following a dispensing error (which was documented as a minor PD). Due to data confidentiality reasons, the results have not been reported for the placebo arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RA101495 0.1 mg/kg (PK) | RA101495 0.3 mg/kg (PK)
Number analyzed (Participants) | 15 | 14
ratio
  RA102758/RA101495- Day 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA102758/RA101495- Day 1: Pre-dose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA102758/RA101495- Day 1: 1 hour postdose: number analyzed (Participants) | 14 | 14
  RA102758/RA101495- Day 1: 1 hour postdose | 0.000 (0.000) | 0.000 (0.000)
  RA102758/RA101495- Day 1: 3 hours postdose | 0.000 (0.000) | 0.000 (0.000)
  RA102758/RA101495- Day 1: 6 hours postdose: number analyzed (Participants) | 14 | 13
  RA102758/RA101495- Day 1: 6 hours postdose | 0.000 (0.000) | 0.013 (0.044)
  RA102758/RA101495- Week 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA102758/RA101495- Week 1: Pre-dose | 0.121 (0.033) | 0.202 (0.038)
  RA102758/RA101495- Week 2: Pre-dose: number analyzed (Participants) | 15 | 13
  RA102758/RA101495- Week 2: Pre-dose | 0.182 (0.038) | 0.307 (0.057)
  RA102758/RA101495- Week 4: Pre-dose: number analyzed (Participants) | 13 | 12
  RA102758/RA101495- Week 4: Pre-dose | 0.197 (0.072) | 0.323 (0.072)
  RA102758/RA101495- Week 8: Pre-dose: number analyzed (Participants) | 15 | 12
  RA102758/RA101495- Week 8: Pre-dose | 0.195 (0.057) | 0.301 (0.070)
  RA102758/RA101495- Week 12: Pre-dose: number analyzed (Participants) | 15 | 13
  RA102758/RA101495- Week 12: Pre-dose | 0.184 (0.065) | 0.303 (0.061)
  RA103488/RA101495- Day 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA103488/RA101495- Day 1: Pre-dose | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ. | NA (NA) — Mean and Standard Deviation are only calculated if at least 2/3 of the individual data points are above LLOQ.
  RA103488/RA101495- Day 1: 1 hour postdose: number analyzed (Participants) | 14 | 14
  RA103488/RA101495- Day 1: 1 hour postdose | 0.000 (0.000) | 0.000 (0.000)
  RA103488/RA101495- Day 1: 3 hours postdose | 0.000 (0.000) | 0.001 (0.001)
  RA103488/RA101495- Day 1: 6 hours postdose: number analyzed (Participants) | 14 | 13
  RA103488/RA101495- Day 1: 6 hours postdose | 0.000 (0.000) | 0.015 (0.045)
  RA103488/RA101495- Week 1: Pre-dose: number analyzed (Participants) | 14 | 14
  RA103488/RA101495- Week 1: Pre-dose | 0.079 (0.037) | 0.099 (0.044)
  RA103488/RA101495- Week 2: Pre-dose: number analyzed (Participants) | 15 | 13
  RA103488/RA101495- Week 2: Pre-dose | 0.104 (0.044) | 0.114 (0.037)
  RA103488/RA101495- Week 4: Pre-dose: number analyzed (Participants) | 13 | 12
  RA103488/RA101495- Week 4: Pre-dose | 0.106 (0.046) | 0.119 (0.038)
  RA103488/RA101495- Week 8: Pre-dose: number analyzed (Participants) | 15 | 12
  RA103488/RA101495- Week 8: Pre-dose | 0.118 (0.044) | 0.127 (0.040)
  RA103488/RA101495- Week 12: Pre-dose: number analyzed (Participants) | 15 | 13
  RA103488/RA101495- Week 12: Pre-dose | 0.116 (0.035) | 0.131 (0.041)

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 122
Description: Treatment emergent adverse events (TEAEs) are defined as an AE that occurs after a treatment start date or an AE that increases in severity after treatment start date. In this study, AEs were planned to be reported for Main portion and Main + Extension portion only.
Groups:
- Main Portion: RA101495 0.1 mg/kg: Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion.
- Main Portion: RA101495 0.3 mg/kg: Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion
- Main Portion: Placebo: Participants received placebo matched to RA101495 as a subcutaneous injection once daily for 12 weeks in the main portion.
- Main and Extension Portion: RA101495 0.1 mg/kg Before Switch to 0.3 mg/kg: Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants who completed main portion and were eligible to enter in the extension period, continued receiving RA101495 0.1 mg/kg up to 48 weeks (until protocol amendment v3.0) in the extension portion.
- Main and Extension Portion: RA101495 0.1 mg/kg After Switch to 0.3 mg/kg: Participants received RA101495 0.1 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. Participants who completed main portion and were eligible to enter in the extension period, continued receiving RA101495 0.1 mg/kg up to Week 48 (until protocol amendment v3.0). Following implementation of protocol amendment v3.0, and upon appropriate reconsent, all study participants ongoing in the extension portion who had previously received the RA101495 0.1mg/kg/day dose switched to receive the RA101495 0.3mg/kg/day until RA101495 is approved and available in the territory, or the sponsor terminates development of RA101495 for gMG. In countries where RA101495 is not approved or marketed, but in which sponsored clinical studies had been conducted, participants received RA101495 through a compassionate use pathway in the extension portion (up to 122 weeks).
- Main and Extension Portion: RA101495 0.3 mg/kg: Participants received RA101495 0.3 mg/kg as a subcutaneous injection once daily for 12 weeks in the main portion. At the end of the treatment period in the main portion, participants received the same dose of study drug in the extension portion until RA101495 is approved and available in the territory, or the sponsor terminates development of RA101495 for gMG. In countries where RA101495 is not approved or marketed, but in which sponsored clinical studies had been conducted, participants received RA101495 through a compassionate use pathway in the extension portion (up to 122 weeks).
Arm/Group | Main Portion: RA101495 0.1 mg/kg | Main Portion: RA101495 0.3 mg/kg | Main Portion: Placebo | Main and Extension Portion: RA101495 0.1 mg/kg Before Switch to 0.3 mg/kg | Main and Extension Portion: RA101495 0.1 mg/kg After Switch to 0.3 mg/kg | Main and Extension Portion: RA101495 0.3 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/15 | 1/22 | 0/21 | 2/21
Serious Adverse Events (participants affected / at risk) | 0/15 | 5/14 | 3/15 | 5/22 | 4/21 | 11/21
Other Adverse Events (participants affected / at risk) | 15/15 | 12/14 | 14/15 | 22/22 | 17/21 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Portion: RA101495 0.1 mg/kg (N=15) | Main Portion: RA101495 0.3 mg/kg (N=14) | Main Portion: Placebo (N=15) | Main and Extension Portion: RA101495 0.1 mg/kg Before Switch to 0.3 mg/kg (N=22) | Main and Extension Portion: RA101495 0.1 mg/kg After Switch to 0.3 mg/kg (N=21) | Main and Extension Portion: RA101495 0.3 mg/kg (N=21)
Worsening of Myasthenia Gravis (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Postoperative hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Portion: RA101495 0.1 mg/kg (N=15) | Main Portion: RA101495 0.3 mg/kg (N=14) | Main Portion: Placebo (N=15) | Main and Extension Portion: RA101495 0.1 mg/kg Before Switch to 0.3 mg/kg (N=22) | Main and Extension Portion: RA101495 0.1 mg/kg After Switch to 0.3 mg/kg (N=21) | Main and Extension Portion: RA101495 0.3 mg/kg (N=21)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 5 (6) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (5)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 3 (3) | 4 (5) | 10 (13) | 3 (4) | 4 (10)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 5 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 2 (2) | 6 (13) | 0 (0) | 3 (3)
Injection site scab (General disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (8)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Worsening of Myasthenia Gravis (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight fluctuation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03315130/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03315130/SAP_001.pdf